CLINICAL TRIAL: NCT05889052
Title: Impact Evaluation of Intermittent Preventive Treatment of Malaria in Infants Plus (IPTi+) in Cameroon: the Plus Project
Brief Title: Perennial Malaria Chemoprevention (PMC) in Cameroon
Status: Active, not recruiting | Type: Observational
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Fobang Institutes Centre for Health Implementation and Translational Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: PLUS-27988-CAM
Record Dates: First submitted 2023-05-03; First posted 2023-06-05 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-10

CONDITIONS: Anemia; Malaria
Keywords: Malaria; Anemia; Perennial Malaria Chemoprevention (PMC); Intermittent Preventative Treatment of Infants (IPTi); Sulfadoxine-pyrimethamine (SP); chemoprevention
MeSH Terms: conditions — Anemia; Malaria | interventions — fanasil, pyrimethamine drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Dried blood spots
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Active cohort control: Children (aged 6-9 months) in the control arm will receive the standard of care: 5 doses of SP at EPI visits (at 10 weeks, 14 weeks, 6 months, 9 months and 15 months).
  Interventions: Drug: Sulfadoxine pyrimethamine
- Active cohort intervention: Children (aged 6-9 months) in the intervention arm with receive PMC: 8 doses of SP at EPI visits (at the same contacts as group 1 plus at 12 months, 18 months and 24 months)
  Interventions: Drug: Sulfadoxine pyrimethamine

INTERVENTIONS:
Drug: Sulfadoxine pyrimethamine — Sulfadoxine-pyrimethamine paediatric formulation (250mg/12.5mg) dispersable tablets (Macleods Pharmaceuticals Ltd)

SUMMARY:
The Plus Project will assess the impact, operational feasibility, efficacy, effectiveness, and cost-effectiveness of PMC. Specifically, the impact evaluation will involve monitoring a passive cohort of all children in the study area reporting all doses of SP received and the number of confirmed cases of malaria and anaemia, as well as a prospective active cohort of children who will have seven home visits over an 18-month period. The total number of participants is expected to be approximately 2,080 children in the areas served by 35 health centres in Cameroon. The results of this study will allow direct evaluation of the protective efficacy of PMC on malaria incidence, severe anaemia, and malaria mortality.

DETAILED DESCRIPTION:
Despite impressive progress in recent years, malaria continues to impose a heavy morbidity and mortality burden. Ninety-five percent of the estimated 247 million malaria cases and 619,000 deaths worldwide in 2021 occurred in the World Health Organization (WHO) Africa Region [1]. The expansion of SP-IPTi to include children up to two years of age and additional entry points, referred to now as PMC, offers the potential to increase the impact of the intervention by delivering more protective doses of SP to an age group with a higher malaria burden. However, to support the development of national policies and international guidelines on the adoption and implementation of PMC at scale, more evidence is needed on where, when, how and under what circumstances PMC can be effective, cost-effective, acceptable, equitable and feasible.

The aim of the impact evaluation is to inform decision-making by policy makers and programme managers involved in national malaria control programmes by evaluating the protective efficacy of PMC with eight doses versus five doses as standard of care in Cameroon. The design is a multi-site quantitative study of the implementation of PMC in Cameroon. The health districts of Soa and Mbankomo were identified as the intervention and control districts, respectively, based on population size, number of Extended Programme of Immunisation (EPI) facilities, malaria incidence, EPI coverage and availability of an appropriate control population receiving standard care.

All children up to 36 months of age with parental consent will be recruited into a passive cohort. The investigators will also extract data on malaria and anaemia cases among children receiving PMC from health facility records.

The investigators will form and follow an active arm of the cohort in which a randomly selected subset of children in the passive cohort will be visited every three months during the study period in their homes to obtain detailed information, including details of the household, malaria risk factors, history of malaria and anaemia, health-seeking behaviour, and past EPI vaccinations. Blood will be collected for microscopy measures of parasitaemia, anaemia diagnosis by haemoglobin levels, and retrospective analysis of malaria infection (not for clinical management) by polymerase chain reaction methods. Rapid diagnostic tests will be used amongst symptomatic children to identify cases. First line antimalarial treatment will be provided to all confirmed cases. Children will be screened for malnutrition by measuring their mid-upper arm circumference (MUAC). If they are determined to have either moderate (MAM) or severe acute malnutrition (SAM), treatment will consist of standard of care which can include referral to the nearest health facility with clinical management capacity or treatment on site.

ELIGIBILITY:
Inclusion Criteria:

* Reside in Soa (intervention) or Mbankomo (control) health districts.
* Agree to take part in the census.
* Aged 6-9 months at the time of enrolment.

Exclusion Criteria:

* Parent/caregiver refused to participate in the cohort.
* Parent/caregiver did not give informed consent.

Max Age: 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children up to 9 months of age in Soa and Mbankomo health districts of Cameroon.
Sampling Method: Probability Sample
Enrollment: 2080 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of malaria infection and clinical malaria | 18 months
  Incidence of: (1) malaria infection, and (2) clinical malaria in children residing in areas designated to receive PMC (intervention) versus standard care (control).

SECONDARY OUTCOMES:
Incidence of severe malaria, malaria deaths, anaemia and severe anaemia | 18 months
  Incidence of: (1) severe malaria, (2) malaria deaths, (3) anaemia, and (4) severe anaemia in children residing in areas designated to receive PMC (intervention) versus standard care (control).
Malaria and anaemia incidence by delivery platform, number of doses and dose schedule | 18 months
  Measure differences in incidence between children residing in areas designated to receive PMC (intervention) versus standard of care (control) based on differences in SP dose patterns by delivery platform, number of doses of SP, and the SP dose schedule.
Dose-response effects of SP on malaria and anaemia | 18 months
  Measure the dose-response effects of SP on incidence of: (1) malaria infection, (2) clinical malaria, (3) severe malaria, (4) anaemia, (5) severe anaemia, and (6) malaria mortality throughout the period of observation.
Effects of distance to health facility on malaria and anaemia | 18 months
  Measure the effects of distance to health facility on incidence of: (1) malaria infection, (2) clinical malaria, (3) severe malaria, (4) anaemia, (5) severe anaemia, and (6) malaria mortality throughout the period of observation.
Incidence of moderate, severe and overall malnutrition | 12 months
  Incidence of: (1) moderate, (2) severe, and (3) overall malnutrition among children residing in areas designated to receive PMC (intervention) versus standard care (control).

CONTACTS AND LOCATIONS:
Overall Officials: Wilfred Mbacham, ScD, Principal Investigator — Fobang Institutes Centre for Health Innovation and Translational Research; R Matthew Chico, MPH, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Multiple, Soa and Mbankomo, Cameroon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] WHO Malaria Report 2022, World Health Organisation
- [Derived] Stresman G, Lal S, Bruce J, Nji A, Serge-Brice A, Mosoff J, McGirr A, Gore-Langton G, McGuire M, Sinsai J, Lele A, Tah-Monunde M, Kouadio ZB, Anatole M, Konate-Toure A, Clarke SE, Gosling R, Mbacham WF, Yavo W, Chico RM. Effectiveness of malaria chemoprevention in the first two years of life in Cameroon and Cote d'Ivoire compared to standard of care: study protocol for a population-based prospective cohort impact evaluation study. BMC Public Health. 2024 Sep 6;24(1):2430. doi: 10.1186/s12889-024-19887-8. PMID 39243075